CLINICAL TRIAL: NCT05000307
Title: Co-Sér: Serological Analysis and Viral Neutralization in People With a Documented COVID-19
Brief Title: Co-Sér: Serological Analysis and Viral Neutralization in People With a Documented COVID-19 Infection
Acronym: Coser
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: BC-08071
Record Dates: First submitted 2021-08-10; First posted 2021-08-11 (Actual); Last update posted 2023-01-11 (Actual); Status verified 2023-01

CONDITIONS: SARS-CoV Infection; Immune System Disorder
Keywords: immunology; SARS-CoV2; Antibodies
MeSH Terms: conditions — Severe Acute Respiratory Syndrome; Immune System Diseases | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: (serial) blood samples in patients with proven SARS-CoV2
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Volunteers, infected with COVID-19 (Experimental)
  Interventions: Diagnostic Test: Blood sample

INTERVENTIONS:
Diagnostic Test: Blood sample — Analysing blood samples for the presence of antibody against SARS-CoV2. When impossible to collect sufficient B-cells for further typing, leucapheresis will be performed if the patient agrees.

SUMMARY:
In light of the current coronavirus disease 2019 (COVID-19) pandemic, the investigators want to better study the immunological characteristics of Severe Acute Respiratory Syndrome-Coronavirus 2 (SARS-CoV2) infections in adults. The investigators invite volunteers to participate in a clinical study to better understand what happens after an infection with SARS-CoV2. By collecting and analysing blood samples of people that were infected, the investigators want to evaluate whether or not the participants had an adaptive immune response with the producting of immunoglobulin. The investigators will evaluate the quality of the antibodies and their neutralising capacity. In a selected patient group with strong antibody response, the investigators will try to reproduce them in the lab after the collection of a larger blood sample (max 72 mL) of, in case of insufficient B-cells, a leucapheresis (after consent of the patient). These antibodies can be used in clinical trials to evaluate whether the investigators can cure patients faster or prevent disease by the utilisation of these antibodies.

Aside from the aforementioned information the investigators will also collect clinical data such as: demographic information, medical history, routine lab results, radiographic imaging and medication use.

After the completion of the study, the samples will be stored for 30 years with consent of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Evidence of prior COVID-19 infection, documented by polymerase chain reaction (PCR) or antibody testing (IgG based)

Exclusion Criteria:

* Known pregnancy at the time of screening
* Patient is on immunosuppressive therapy or was treated with immunosuppressive therapy during the last 6 months
* Inability to give informed consent or absence of legal representative who can give informed consent.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 79 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-01-27 (Actual)

PRIMARY OUTCOMES:
Neutralising capacity of naturally produced antibodies against SARS-CoV2 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Linos Vandekerckhove, MD PhD, Principal Investigator — PI
Locations (1):
- Ghent University Hospital, Ghent, Oost-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: No